CLINICAL TRIAL: NCT01226069
Title: To Investigate the Effectiveness of Topical Glycerine Sulphate, Hirudoid Cream and Nil Application in Treating Peripheral Cannula Related Phlebitis
Brief Title: Effectiveness of Topical Glycerine Sulphate Paste, Hirudoid Cream and Nil Application on Superficial Phlebitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Isabel Ng Hui Leng, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D/09/481
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Infection
Keywords: superficial phlebitis; cannula-related vein inflammation; Glycerine magnesium sulphate; Hirudoid cream; Nursing
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glycerine Magnesium Sulphate paste (Active Comparator)
  Interventions: Drug: Glycerine Magnesium sulphate paste
- Hirudoid cream (Active Comparator): Topical Mucopolysaccharide polysulphate
  Interventions: Drug: Mucopolysaccharide polysulphate
- No application (Experimental): Patient will not receive any topical application to apply on the phlebitis site. The outcome assessor will monitor regularly at pre-determined schedule as patients in other active arms.
  Interventions: Other: No application

INTERVENTIONS:
Drug: Glycerine Magnesium sulphate paste — Dosage to apply adheres to the manufacturer's recommendation. Sufficient amount should cover the erythema size. Dose frequency is 12 hourly.
  Arms: Glycerine Magnesium Sulphate paste
Drug: Mucopolysaccharide polysulphate — Dosage to apply adheres to the manufacturer's recommendation. Sufficient amount should cover the erythema size. Dose frequency is 12 hourly.
  Arms: Hirudoid cream
Other: No application — No application
  Arms: No application

SUMMARY:
The aim of the interventional study is to compare the different treatment modalities in reducing erythema size and rate of resolving phlebitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the study institution between Dec 2009 and Feb 2010 and observed to develop redness associated with peripheral infusion cannula.

Exclusion Criteria:

* Thrombosis, poor skin condition, and pus seen at the previous puncture.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Erythema size | 5 days
  The incremental percentage change in erythema size

SECONDARY OUTCOMES:
Time to resolve redness | 5 days
  The rate of phlebitis resolution

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Ng, MSc Epidemiology, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Result] dos Reis PE, Silveira RC, Vasques CI, de Carvalho EC. Pharmacological interventions to treat phlebitis: systematic review. J Infus Nurs. 2009 Mar-Apr;32(2):74-9. doi: 10.1097/NAN.0b013e318198d497. PMID 19289920
- [Result] Almenar L, Hernandez M, Gimeno JV, Palencia M, Algarra F. [Heparinoids versus nitroglycerin in the treatment of superficial phlebitis]. Rev Clin Esp. 1993 Oct;193(5):229-31. Spanish. PMID 8256008
- [Result] Cokmez A, Gur S, Genc H, Deniz S, Tarcan E. Effect of transdermal glyceryl trinitrate and anti-inflammatory gel in infusion phlebitis. ANZ J Surg. 2003 Oct;73(10):794-6. doi: 10.1046/j.1445-2197.2003.02791.x. PMID 14525568
- [Result] Gouping Z, Wan-Er T, Xue-Ling W, Min-Qian X, Kun F, Turale S, Fisher JW. Notoginseny cream in the treatment of phlebitis. J Infus Nurs. 2003 Jan-Feb;26(1):49-54. doi: 10.1097/00129804-200301000-00007. PMID 12544367
- [Result] Vilardell M, Sabat D, Arnaiz JA, Bleda MJ, Castel JM, Laporte JR, Vallve C. Topical heparin for the treatment of acute superficial phlebitis secondary to indwelling intravenous catheter. A double-blind, randomized, placebo-controlled trial. Eur J Clin Pharmacol. 1999 Feb;54(12):917-21. doi: 10.1007/s002280050575. PMID 10192751
- [Result] Gua H, Li Y-J, Ma H-J. Efficacy observation of glycerine magnesium sulphate emulsion on the treatment of phlebitis. Journal of Lanzhou University (Medical Sciences). 2007;33(2):67-69.